CLINICAL TRIAL: NCT04536285
Title: Clinical Characteristics and Outcome of Hospitalized Children and Adolescent Patients With Type 1 Diabetes During the COVID-19 Pandemic: Data From a Single Center Surveillance Study in Egypt
Brief Title: Hospitalized Children and Adolescent Patients With Type 1 Diabetes During the COVID-19 Pandemic in Egypt
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Eman Monir Sherif, Professor of Pediatrics, Ain Shams University
Other Study IDs: FMASU P59/2020
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Type 1 Diabetes; Covid19
Keywords: Type 1 Diabetes; Covid 19; Diabetic ketoacidosis
MeSH Terms: conditions — Diabetes Mellitus, Type 1; COVID-19; Diabetic Ketoacidosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although reports showed that children with well controlled diabetes do not appear to have increased risk of infection with SARS-CoV-2, however data are scarce regarding the extent to which clinical and demographic data of patient could modify the outcome and severity of the disease. Additionally, the link between covid-19 and diabetes remains controversial.

DETAILED DESCRIPTION:
Data from poorly controlled patients with type 1 diabetes remains controversial regarding whether diabetes itself could increases the susceptibility of infection with SARS-CoV-2 and subsequently impacts the outcomes in these patients , or the SARS-CoV-2 subsequently affects the risk of type 1 diabetes and increase in the prevalence of severe DKA.

Poorly controlled diabetes and chronic hyperglycemia creates a state of low grade chronic inflammation, which may explain the underlying mechanism of increased susceptibility to infection and infer the outcome in patients with diabetes .

Poorly controlled diabetes has been linked to multiple derangements of immune system including inhibition of lymphocyte proliferation in response to different stimuli, as well as impaired monocyte/macrophage function together with increased synthesis of pro-inflammatory cytokines and adhesion molecules that mediate tissue inflammation .

Few data links the association between development of diabetic ketoacidosis in patients with COVID-19, where the infection could trigger higher stressful conditions, with the release of stress hormones leading to increased blood glucose levels and abnormal glucose variability .

The extent to which clinical and demographic data of patients with type 1 diabetes modifies the outcome and severity of the disease seems entirely unclear and is the question of several researches.

• Study Tools:

All patients admitted to Pediatrics Hospital, Ain Shams University in the period between May to August 2020 will be subjected to:

1- Detailed history 2. Thorough clinical examination: To assess the inclusion and exclusion criteria. A thorough clinical review to assess organ involvements and clinical and laboratory characteristics as well as the outcome measures in the studied cohort.

3. Data collection: Demographic and data will be extracted from patients inpatient files and reports

ELIGIBILITY:
Inclusion Criteria:

* All patients with type 1 diabetes admitted to Pediatrics Hospital, Ain Shams University in the period between May to July 2020.
* Age: less than 18 years old.

Exclusion Criteria:

• Children with other forms of diabetes, including: type 2, monogenic forms and secondary diabetes

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All diabetic patients admitted to Pediatrics Hospital, Ain Shams University in the period between May to August 2020.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Clinical characteristic of pediatric and adolescent patients with type 1 diabetes hospitalized with COVID -19. | 4 months
  complications and comorbidities associated with diabetes
Laboratory characteristic of pediatric and adolescent patients with type 1 diabetes hospitalized with COVID -19. | 4 months
  Acute phase reactants
Prognosis of pediatric and adolescent patients with type 1 diabetes hospitalized with COVID -19. | 4 month
  Intensive care admission

SECONDARY OUTCOMES:
Incidence of new onset type 1 diabetes among confirmed cases of Covid-19 infection among children and adolescents | 4 months
  Incidence of new onset type 1 diabetes among confirmed cases of Covid-19 infection among children and adolescents
Presentation of diabetes and its acute complications among pediatric and adolescent patients with type 1 diabetes during COVID-19 Pandemic in Egypt | 4 month
  Impact of Covid-19 pandemic on presentation of diabetes and its acute complications among pediatric and adolescent patients with type 1 diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Yasmine Elhenawy, Study Director — Ain Shams University
Locations (1):
- Pediatrics and Adolescents Diabetes Unit (PADU), Pediatrics Hospital, Faculty of Medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided